CLINICAL TRIAL: NCT00259974
Title: Double-blind Randomized Trial of Rituximab Versus Placebo in Polyneuropathy Associated With Anti-MAG IgM Monoclonal Gammopathy
Brief Title: RIMAG Study: Trial of Rituximab Versus Placebo in Polyneuropathy Associated With Anti-MAG IgM Monoclonal Gammopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Bordeaux (Other); University Hospital, Limoges (Other); Henri Mondor University Hospital (Other); University Hospital, Marseille (Other); Hospices Civils de Lyon (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Isabelle BRINDEL, Department of Clinical Research of developpement
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P040409
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2007-03

CONDITIONS: Polyneuropathy
Keywords: Anti-MAG monoclonal gammopathy; Polyneuropathy; Rituximab
MeSH Terms: conditions — Polyneuropathies | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab

SUMMARY:
Polyneuropathy associated with anti-MAG monoclonal IgM gammopathy is responsive of mainly a sensory deficit in predominantly males ,aged 40-70 years. Significantly high serum anti-MAG antibodies are linked with demyelinating features of the peripheral nerves.Rituximab, an anti-CD 20 monoclonal antibody is a new drug which reduces B-lymphocytes. This study will test the safety and efficacy of rituximab in the treatment of patients with anti-MAG polyneuropathy.

DETAILED DESCRIPTION:
Acting of a polyneuropathy for which there is not any treatment of reference today (see supra), a test of double-knowledge versus placebo is justified. Acting of a chronic polyneuropathy, the clinical evaluation must be led over one one year period. Acting of a sensitive polyneuropathy and the awaited benefit being the IMPROVEMENT OF the CLINICAL SIGNS, the principal criterion is a sensitive score in addition validated in chronic sensitive polyneuropathies immunodeficiency syndrome.

The patients answering the criteria of inclusion and none inclusion (see V-2) will be randomized in 2 groups: the first group will receive a perfusion IV of rituximab to the amount of 375 mg/m2 of body surface, once per week, during 4 weeks (see VII-3); the second group will receive 4 perfusions IV of placebo according to same methods'. The evaluation (see VI-1) will be carried out at the time of the randomization, then repeated in 3 months, 6 months, 9 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* IgM monoclonal gammopathy
* Anti-MAG antibody titers > 1.1000 BTU (ELISA)
* Worsening polyneuropathy with INCAT score > 4
* Informed consent

Exclusion Criteria:

* Severe comorbidity
* Other concurrent causes of polyneuropathy
* Concurrent immunosuppressive therapies (wash-out > 3 months)
* Previous treatment with rituximab
* Lymphoproliferative disease indicating other immunosuppressive treatment
* Unability to follow-up
* Previous documented side-effects with components involved in the tested drug
* White cell count < 1500/mm3 or platelet count < 75.000/mm3
* Patient under law

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
INCAT sensory score at 1 year | during de study
  INCAT sensory score at 1 year

SECONDARY OUTCOMES:
Functional scales, MRC score | during the study
  Functional scales, MRC score
Quality of life (SF 36) | during the study
  Quality of life (SF 36)
Serum lymphocytes count, IgM level, anti-MAG antibody titers | during the study
  Serum lymphocytes count, IgM level, anti-MAG antibody titers
Electrophysiological parameters | during the study
  Electrophysiological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc LEGER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Consultation de Pathologie Neuromusculaire, Bâtiment Babinski, Paris, France

REFERENCES:
- [Background] Leger JM. A review of the medical management of chronic inflammatory demyelinating polyradiculoneuropathy. Expert Opin Pharmacother. 2005 Apr;6(4):569-82. doi: 10.1517/14656566.6.4.569. PMID 15934883